CLINICAL TRIAL: NCT02544854
Title: Pharmacokinetic/Pharmacodynamic Model of Propofol in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 15-068
Record Dates: First submitted 2015-09-06; First posted 2015-09-09 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia
Keywords: Pharmacokinetics, pharmacodynamics, propofol, pediatrics
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ages 1 year - 3 years 11 months (Experimental): Propofol infusion, measuring of plasmatic levels of propofol through venous sampling
  Interventions: Drug: Propofol
- Ages 4 years - 8 years 11 months (Experimental): Propofol infusion, measuring of plasmatic levels of propofol through venous sampling
  Interventions: Drug: Propofol
- Ages 9 years - 11 years 11 months (Experimental): Propofol infusion, measuring of plasmatic levels of propofol through venous sampling
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol infusion will be started after inhalational induction by manual infusion by the following scheme:
  1. First 15 minutes: 15 mg/kg/min
  2. 16 to 30 minutes: 13 mg/kg/min
  3. 31 to 60 minutes: 11 mg/kg/min
  4. 61 to 120 minutes: 10 mg/kg/min Dose will be titrated to maintain BIS between 40 - 50.
  Venous sampling for plasmatic levels of propofol measuring will be made at the following moments:
  1. 5, 15 and 25 minutes of starting infusion,
  2. 1, 3, 5, 7, 9 and 12 minutes of bolus and,
  3. 5, 25, 60 and 120 minutes of infusion ended.
  Other Names: Diprivan

SUMMARY:
By measuring plasmatic concentration of propofol at different intervals during surgery of children aged 1 to 12 years old and measuring Bispectral Index (BIS) as a surrogate for cerebral activity, the investigators aim to create a pharmacokinetic/pharmacodynamic model of propofol for children.

DETAILED DESCRIPTION:
Propofol is an intravenous anesthetic capable of providing a safe general anesthesia, free from many of the adverse effects associated with inhalation anesthetics (postoperative nausea and vomiting, agitation on awakening, seizures and trigger malignant hyperthermia crisis) and widely used in adults, but even less so in children. This is due to the fact that its pharmacological characteristics have not been clarified at all in the pediatric population.

The physiological maturation of different systems in children, as well as changes in body composition and metabolism may determine significant changes in the pharmacokinetics (distribution volumes and clearance) of children. Moreover, within the same age group, variations across different individuals may make even less predictable the pharmacokinetic models currently in use. Indeed, previous work in our group based on these models have shown that propofol dosage required by children to induce general anesthesia is inversely proportional to the age, which could be explained by biases in these models, different sensitivity to propofol at different ages and sizes, etc.

The effect of propofol in the brain is described by its pharmacodynamics, but in children this is still in debate. Using a brain activity monitor (BIS), the effect of propofol at the central nervous system can be analyzed under a model of nonlinear mixed effects (NONMEM) and establish the time to peak effect to characterize in detail the pharmacodynamics of this drug.

Integrating pharmacokinetic and pharmacodynamic data, a pharmacokinetic/pharmacodynamic (PK/PD) model for the pediatric population can be derived.

The aim of this paper is to describe the first PK / PD model of propofol in children, valid for different ages and to analyze them in the context of different body composition parameters.

The importance of this study is that its results will publish the missing link in the pediatric pharmacology of propofol, which will encourage more research and more widespread use of this technique in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 year through 11 years 11 months and 29 days old.
* American Society of Anesthesiology (ASA) score 1 or 2.
* Elective surgery of more than 1 hour of expected duration.
* Written informed consent signed by parents or legal guardians.
* Oral and written consent in children aged over 7 years old.

Exclusion Criteria:

* Known allergies to study drugs.
* Use of any medication acting on central nervous system in the last 24 hours previous to surgery.
* Chronic cardiac, renal, hepatic or neurologic disease that determines abnormal function.
* Difficult airway (predicted or known).
* Use of neuraxial anesthesia.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Propofol plasmatic levels | From start of infusion: 5 min, 15 min, 45 min; from bolus 0 min, 1 min, 3 min, 5 min, 10 min; after infusion 30 min, 60 min, 120 min, 360 min
  Measured by high pressure liquid chromatography

SECONDARY OUTCOMES:
Hemodynamics | Entering operating room up to end of anesthesia
  Heart rate and arterial pressure
Propofol total dose | Start of propofol infusion until it ends
  Measured in milligrams
Sevoflurane total dose | Start of inhalational induction to zero end tidal concentration
Pulse oximetry | Entering operating room up to end of anesthesia
BIS | Entering operating room up to end of anesthesia
  Depth of anesthesia will be recorded with BIS monitor

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Fuentes, MD, Principal Investigator — Professor; Rose M Heider, MD, Principal Investigator — Professor
Locations (1):
- Division de Anestesia - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gibert S, Sabourdin N, Louvet N, Moutard ML, Piat V, Guye ML, Rigouzzo A, Constant I. Epileptogenic effect of sevoflurane: determination of the minimal alveolar concentration of sevoflurane associated with major epileptoid signs in children. Anesthesiology. 2012 Dec;117(6):1253-61. doi: 10.1097/ALN.0b013e318273e272. PMID 23103557
- [Background] Kearns GL, Reed MD. Clinical pharmacokinetics in infants and children. A reappraisal. Clin Pharmacokinet. 1989;17 Suppl 1:29-67. doi: 10.2165/00003088-198900171-00005. PMID 2692939
- [Background] Fuentes R, Cortinez I, Ibacache M, Concha M, Munoz H. Propofol concentration to induce general anesthesia in children aged 3-11 years with the Kataria effect-site model. Paediatr Anaesth. 2015 Jun;25(6):554-9. doi: 10.1111/pan.12657. Epub 2015 Apr 16. PMID 25880448
- [Background] Rigouzzo A, Servin F, Constant I. Pharmacokinetic-pharmacodynamic modeling of propofol in children. Anesthesiology. 2010 Aug;113(2):343-52. doi: 10.1097/ALN.0b013e3181e4f4ca. PMID 20613468
- [Background] Coppens MJ, Eleveld DJ, Proost JH, Marks LA, Van Bocxlaer JF, Vereecke H, Absalom AR, Struys MM. An evaluation of using population pharmacokinetic models to estimate pharmacodynamic parameters for propofol and bispectral index in children. Anesthesiology. 2011 Jul;115(1):83-93. doi: 10.1097/ALN.0b013e31821a8d80. PMID 21555936
- [Background] Panchatsharam S, Callaghan M, Day R, Sury MR. Measured versus predicted blood propofol concentrations in children during scoliosis surgery. Anesth Analg. 2014 Nov;119(5):1150-7. doi: 10.1213/ANE.0000000000000413. PMID 25225889
- [Background] Howie SR. Blood sample volumes in child health research: review of safe limits. Bull World Health Organ. 2011 Jan 1;89(1):46-53. doi: 10.2471/BLT.10.080010. Epub 2010 Sep 10. PMID 21346890
- [Derived] Fuentes R, Cortinez LI, Contreras V, Ibacache M, Anderson BJ. Propofol pharmacokinetic and pharmacodynamic profile and its electroencephalographic interaction with remifentanil in children. Paediatr Anaesth. 2018 Dec;28(12):1078-1086. doi: 10.1111/pan.13486. Epub 2018 Oct 11. PMID 30307663